CLINICAL TRIAL: NCT04174807
Title: Prospective Study of Antenatal Diagnostic Criteria for Digestive Complications of Gastroschisis
Acronym: LaparoDAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49-RC18-0155
Record Dates: First submitted 2019-11-05; First posted 2019-11-22 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Gastroschisis; Intestinal Occlusion
Keywords: gastroschisis; prenatal diagnosis; gastrointestinal complications; wall defect; predictive factors
MeSH Terms: conditions — Gastroschisis; Intestinal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
Gastroschisis is a rare congenital malformation consisting in a right para-umbilical defect of the abdominal wall leading to an evisceration of the abdominal content. About 25% of the cases are associated with intestinal malformation, leading to an increase in peri-natal morbidity and mortality. No prospective study has been able to definitely describe predictive factors for complicated gastroschisis on prenatal ultrasound examinations.

The aim of the current study is to prospectively look for US prenatal features predictive of complicated gastroschisis, on a national multicentric cohort.

Patients will be included during the 22 weeks of amenorrhea (WA) ultrasound examination, and pre- and postnatal clinical data will be recorded up to the 6th months of the child.

Data will then be analysed and compared in the groups of simple or complicated gastroschisis, in order to define pre-natal prognostic factors, to correlate them with specific prognosis, and to might better determine specific strategies for better care of these patients.

ELIGIBILITY:
Inclusion Criteria:

Every volunteer pregnant woman, in whom an antenatal ultrasound diagnosis of gastroschisis has been carried, before the end of 22 weeks of amenorrhea.

Exclusion Criteria:

Lack of informed consent or refusal of the person to participate in study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women diagnosed with gastroschisis in antenatal and newborns diagnosed with gastroschisis from birth to 6 months of life.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the collar diameter/abdominal circumference ratio as a predictive factor of complex gastroschisis. | 2,5 years
  The measures of the collar diameter/abdominal circumference ratio on antenatal ultrasound examination will be evaluated as predictive factor of complex gastroschisis

SECONDARY OUTCOMES:
Evaluation of antenatal ultrasound in predictive diagnosis of complex gastroschisis | 2,5 years
  Identify other predictive ultrasound factors of complex gastroschisis among the different ultrasound measurements, such as gastric dilatation, maximum diameter of the intraabdominal loop, ...
Composite predictive criterion of complex gastroschisis | 2,5 years
  Define the existence of a composite predictive criterion of complex gastroschisis that incorporates all or several predictive ultrasound factors
Composite predictive criterion of complex gastroschisis by MRI | 2,5 years
  Perform the same measurements as for outcome 3 by MRI
Research risk factors in the mother | 2,5 years
  Search for risk factors for complex gastroschisis from medical examination of the mother (age, tobacco, drugs, body mass index, exposure to chemicals)
Propose a decision algorithm for prenatal management of these patients | 2,5 years
  Based on identified risk factors
Measure the impact of complex gastroschisis on follow-up until 6 months of children | 6 months of child's life
  Use of different parameters (clinical assessment at 6 months, medical history) to evaluate the impact of complex gastroschisis on children at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Françoise SCHMITT, Dr, Principal Investigator — UH Angers
Locations (36):
- France (35):
  - University Hospital of Amiens, Amiens
  - University Hospital of Angers, Angers
  - University Hospital of Besançon, Besançon
  - University Hospital of Bordeaux, Bordeaux
  - University Hospital of Brest, Brest
  - University Hospital of Caen, Caen
  - University Hospital of Bicêtre, Clamart
  - University Hospital of Clermont-Ferrand, Clermont-Ferrand
  - University Hospital of Dijon, Dijon
  - University Hospital of Grenoble, Grenoble
  - University Hospital of Le Havre, Le Havre
  - University Hospital of Le Mans, Le Mans
  - University Hospital of Lens, Lens
  - University Hospital of Lille, Lille
  - University Hospital of Limoges, Limoges
  - University Hospital of Lyon, Lyon
  - University Hospital of Marseille, Marseille
  - University Hospital of Montpellier, Montpellier
  - University Hospital of Nancy, Nancy
  - University Hospital of Nantes, Nantes
  - University Hospital of Nice, Nice
  - University Hospital of Nîmes, Nîmes
  - University Hospital of Orléans, Orléans
  - University Hospital of Necker, Paris
  - University Hospital of Robert Debré, Paris
  - University Hospital of Trousseau, Paris
  - University Hospital of Poitiers, Poitiers
  - University Hospital of René Dubos, Pontoise
  - University Hospital of Reims, Reims
  - University Hospital of Rennes, Rennes
  - University Hospital of Rouen, Rouen
  - University Hospital of Saint-Etienne, Saint-Etienne
  - University Hospital of Strasbourg, Strasbourg
  - University Hospital of Toulouse, Toulouse
  - University Hospital of Tours, Tours
- University Hospital of Fort de France, Fort-de-France, Martinique

REFERENCES:
- [Result] Geslin D, Clermidi P, Gatibelza ME, Boussion F, Saliou AH, Le Manac'h Dove G, Margaryan M, De Vries P, Sentilhes L, Levard G, Lardy H, Arnaud A, Leclair MD, Podevin G, Schmitt F. What prenatal ultrasound features are predictable of complex or vanishing gastroschisis? A retrospective study. Prenat Diagn. 2017 Feb;37(2):168-175. doi: 10.1002/pd.4984. Epub 2017 Jan 25. PMID 27981591
- [Result] Kassa AM, Lilja HE. Predictors of postnatal outcome in neonates with gastroschisis. J Pediatr Surg. 2011 Nov;46(11):2108-14. doi: 10.1016/j.jpedsurg.2011.07.012. PMID 22075340
- [Result] Kuleva M, Khen-Dunlop N, Dumez Y, Ville Y, Salomon LJ. Is complex gastroschisis predictable by prenatal ultrasound? BJOG. 2012 Jan;119(1):102-9. doi: 10.1111/j.1471-0528.2011.03183.x. Epub 2011 Oct 21. PMID 22017923